CLINICAL TRIAL: NCT01114984
Title: A Prospective Cohort Study to Evaluate the Incidence and Characteristics of Post-Operative Pain Among Patients Undergoing Various Breast Surgeries
Brief Title: Post-Breast Procedure Pain Syndrome Study
Status: Withdrawn | Type: Observational
Why Stopped: Bad design.
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Roya Yumul, M.D.,PhD., Residency program director, Department of anesthesiology, Cedars-Sinai Medical Center
Other Study IDs: Pro00019341
Record Dates: First submitted 2010-04-23; First posted 2010-05-03 (Estimated); Last update posted 2015-03-02 (Estimated); Status verified 2015-02

CONDITIONS: Breast; Mastectomy, Segmental
Keywords: Pain management; Radical mastectomy; Breast surgery; post-operative pain
MeSH Terms: conditions — Agnosia; Pain, Postoperative

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (8):
- 10% after breast biopsy: Incidence Post-operative pain after breast surgery.
- 20% after lumpectomy: Incidence Post-operative pain after breast surgery
- 30% after simple mastectomy: Incidence Post-operative pain after breast surgery
- 50% after mastectomy with reconstruction: Incidence Post-operative pain after breast surgery
- 50% after radical mastectomy: Incidence Post-operative pain after breast surgery
- 50% after radi mastectomy+reconstruction: Incidence Post-operative pain after breast surgery after radical mastectomy with reconstruction
- 40% after cosmetic augmentation: Incidence Post-operative pain after breast surgery
- 40% after breast reduction: Incidence Post-operative pain after breast surgery

SUMMARY:
The purpose of this study is to better understand and characterize the pain that some patients experience after undergoing various breast surgeries, including breast biopsy, lumpectomy, mastectomy, mastectomy with reconstruction, cosmetic breast augmentation, and breast reduction.

DETAILED DESCRIPTION:
Post-operative breast pain is one of the most common adverse effects after breast surgery procedures. According to previous studies, anywhere from 20-60% of breast surgery patients report mastalgia as an adverse outcome of surgery (1, 2). Although the exact mechanism has not been well defined, the pain is generally neuropathic in nature and described as a burning sensation, electric and shock like, with a stabbing quality (2,3). The large majority of post-operative mastalgia is therefore believed to be secondary to nerve damage, particularly injury to the intercostobrachial nerve, and less commonly the long thoracic, medial and lateral pectoral, and/or the thoracodorsal nerves. Other reported causes of post-operative breast pain include scarring pain, lymphedema, radiation plexopathy, and hematomas (1-5).

Increasing rates of breast surgeries, whether elective, diagnostic, prophylactic, or therapeutic, warrant a more detailed examination of this pain-syndrome, particularly as previous research in the area is rather limited and narrow. A better understanding of the potential mechanisms causing pain, as well as more accurate and current incidence rates, and comparisons of adverse outcomes among the various options available to patients can help guide physicians towards improved clinical practices and patients towards more informed decision-making. Therefore, we designed this prospective cohort study to better understand the underlying mechanisms which may cause post-operative pain after various types of breast surgeries including breast biopsy, lumpectomy, mastectomy, mastectomy with reconstruction, cosmetic augmentation, and breast reduction, as well as to compare and contrast incidence, quality, and distribution of the post-operative pain caused by these various surgical procedures.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo one or more of the breast surgical procedures being studied for this project
* Willingness and ability to sign an informed consent document
* No allergies to anesthetic or analgesic medications
* Female,
* 18-80 years of age
* ASA class I-III adult

Exclusion Criteria:

* Patients with known allergy, hypersensitivity or contraindications to anesthetic or analgesic medications
* Patients with clinically-significant medical conditions, such as brain, heart, kidney, endocrine, or liver diseases, or history of chronic pain syndrome or neuropathy.
* Subjects with a history of alcohol or drug abuse within the past 3 months
* Subjects with a history of pain medication abuse
* Any other conditions or use of any medication which may interfere with the conduct of the study

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergo breast surgery. (breast biopsy, lumpectomy, simple mastectomy,mastectomy with reconstruction, radical mastectomy, radical mastectomy with reconstruction, cosmetic augmentation and breast reduction)
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2009-07; Primary Completion 2014-06 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Postoperative Pain using VRS | 6 months
  prospective cohort evaluation of patients undergoing various breast surgery procedures, followed for a period of 6 months post-operatively, and assessed for post-operative breast pain.

SECONDARY OUTCOMES:
Opioid consumption obtained from the recorded data | 6 months
  Perioperative use of opioid consumption inside hospital (recorded by study staff and data obtained from patient charts) Post discharge use of opioid consumption (data obtained from the follow up questionnaires at 1, 2, or 3, then 7 days and at 6 months after surgery)
Postoperative nausea and vomiting using a Verbal Rating Scale | 6 months
  Outcomes will be measured with follow up questionnaires at 1, 2, or 3, then 7 days and 6 months after surgery
Return to normal activities of daily living using follow up questionnaires | 6 months
  Questionnaires will help evaluate patients recovery and return to normal activities of daily living(including dietary intake, bowel and bladder function, physical activities). Patients will be contacted via mail or e-mail.
Patient satisfaction using a verbal rating scale from 0 to 100 | 6 months
  Patients will state their satisfaction level on a scale of 0= Not satisfied to 100= Excellent
Hospital stay | up to 1 week
  Record number of days patients remain in hospital

CONTACTS AND LOCATIONS:
Overall Officials: Roya Yumul, MD, PhD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars Sinai Medical Center, Los Angeles, California, United States